CLINICAL TRIAL: NCT00853671
Title: Myocardial Stress Perfusion Imaging With Dual Source CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Brian Burns Ghoshhajra, Clinical Director, Cardiac CT and MRI, Department of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSCTSTRESS
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Multidetector Computed Tomography; Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine; Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adenosine Stress Dual-source CTP (Experimental): A multiphase adenosine Stress Dual-source stress perfusion computed tomography imaging test, as described above, will be performed in all patients.
  Interventions: Other: Adenosine Stress Dual-source CTP

INTERVENTIONS:
Other: Adenosine Stress Dual-source CTP — Adenosine- continuous infusion at 140mcg/ kg/ min for 2.5 min; Iopamidol (IV contrast)- total dose of 150cc; Siemens SOMATOM Definition CT scanner (CT scan radiation) - effective radiation dose of approximately 13mSv (tube voltage 120kV, tube current 340mAs for one retrospectively gated cardiac CT with tube current modulation and two prospectively gated cardiac CTs on a Dual Source scanner)
  This is an observational trial, and all patients will undergo the Adenosine Stress Dual-source CTP procedure.
  Other Names: Adenosine; Iopamidol 370; Siemens SOMATOM Definition

SUMMARY:
The investigators propose a novel technique using dual source multidetector computed tomography (DSCT) where information on both coronary anatomy and myocardial perfusion is obtained in a single scan. The investigators hypothesize that a coronary CTA protocol can be devised to obtain resting myocardial perfusion, myocardial perfusion after stress, and coronary anatomy. Hence, one diagnostic test will be able to detect the presence of coronary plaque as well as assess the functional significance of a stenosis.

ELIGIBILITY:
Inclusion Criteria:

* A prior adenosine or exercise stress SPECT exam with high likelihood of being referred to the cardiac catheterization laboratory for invasive angiogram
* Age > 40 years old
* Able to comprehend and sign the consent form.

Exclusion Criteria:

* Acute coronary syndromes (unstable angina, non-ST elevation myocardial infarction, ST elevation myocardial infarction)
* Unstable clinical conditions (i.e. hemodynamic instability, arrhythmias)
* Premenopausal women who have a positive pregnancy test.
* Serum Creatinine level ≥1.5 mg/dl as an indicator of renal insufficiency.
* Known allergy to iodinated contrast agents
* Atrial fibrillation
* Asthma
* Critical aortic stenosis
* Systolic blood pressure < 90 mmHg
* Advanced heart block

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian B Ghoshhajra, MD, Principal Investigator — Massachusetts General Hospital; Ricardo C Cury, MD, Study Director — Massachusetts General Hospital, Baptist Hospital, Miami
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hulten EA, Bittencourt MS, Ghoshhajra B, Blankstein R. Stress CT perfusion: coupling coronary anatomy with physiology. J Nucl Cardiol. 2012 Jun;19(3):588-600. doi: 10.1007/s12350-012-9546-5. PMID 22456969
- [Background] Techasith T, Cury RC. Stress myocardial CT perfusion: an update and future perspective. JACC Cardiovasc Imaging. 2011 Aug;4(8):905-16. doi: 10.1016/j.jcmg.2011.04.017. PMID 21835384
- [Result] Blankstein R, Shturman LD, Rogers IS, Rocha-Filho JA, Okada DR, Sarwar A, Soni AV, Bezerra H, Ghoshhajra BB, Petranovic M, Loureiro R, Feuchtner G, Gewirtz H, Hoffmann U, Mamuya WS, Brady TJ, Cury RC. Adenosine-induced stress myocardial perfusion imaging using dual-source cardiac computed tomography. J Am Coll Cardiol. 2009 Sep 15;54(12):1072-84. doi: 10.1016/j.jacc.2009.06.014. PMID 19744616
- [Result] Rocha-Filho JA, Blankstein R, Shturman LD, Bezerra HG, Okada DR, Rogers IS, Ghoshhajra B, Hoffmann U, Feuchtner G, Mamuya WS, Brady TJ, Cury RC. Incremental value of adenosine-induced stress myocardial perfusion imaging with dual-source CT at cardiac CT angiography. Radiology. 2010 Feb;254(2):410-9. doi: 10.1148/radiol.09091014. PMID 20093513
- [Result] Okada DR, Ghoshhajra BB, Blankstein R, Rocha-Filho JA, Shturman LD, Rogers IS, Bezerra HG, Sarwar A, Gewirtz H, Hoffmann U, Mamuya WS, Brady TJ, Cury RC. Direct comparison of rest and adenosine stress myocardial perfusion CT with rest and stress SPECT. J Nucl Cardiol. 2010 Jan-Feb;17(1):27-37. doi: 10.1007/s12350-009-9156-z. PMID 19936863
- [Result] Uthamalingam S, Gurm GS, Sidhu MS, Verdini DJ, Vorasettakarnkij Y, Engel LC, Blankstein R, Mamuya WS, Hoffman U, Brady TJ, Cury RC, Ghoshhajra BB. Comparison of dual-source 64-slice adenosine stress CT perfusion with stress-gated SPECT-MPI for evaluation of left ventricular function and volumes. J Cardiovasc Comput Tomogr. 2012 Jan-Feb;6(1):24-30. doi: 10.1016/j.jcct.2011.10.016. Epub 2011 Nov 18. PMID 22222164
- [Result] Ghoshhajra BB, Maurovich-Horvat P, Techasith T, Medina HM, Verdini D, Sidhu MS, Blankstein R, Brady TJ, Cury RC. Infarct detection with a comprehensive cardiac CT protocol. J Cardiovasc Comput Tomogr. 2012 Jan-Feb;6(1):14-23. doi: 10.1016/j.jcct.2011.10.014. Epub 2011 Nov 18. PMID 22210535
- [Result] Ghoshhajra BB, Rogers IS, Maurovich-Horvat P, Techasith T, Verdini D, Sidhu MS, Drzezga NK, Medina HM, Blankstein R, Brady TJ, Cury RC. A comparison of reconstruction and viewing parameters on image quality and accuracy of stress myocardial CT perfusion. J Cardiovasc Comput Tomogr. 2011 Nov-Dec;5(6):459-66. doi: 10.1016/j.jcct.2011.10.011. Epub 2011 Oct 31. PMID 22146505

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 3/3/2008 - 7/1/2009
Groups:
- Myocardial Stress CT Perfusion Imaging: Patients who will undergo myocardial stress CT perfusion imaging. Adenosine- continuous infusion at 140mcg/ kg/ min for 2.5 min; Iopamidol (IV contrast)- total dose of 150cc; Siemens SOMATOM Definition CT scanner (CT scan radiation) - effective radiation dose of approximately 13mSv (tube voltage 120kV, tube current 340mAs for one retrospectively gated cardiac CT with tube current modulation and two prospectively gated cardiac CTs on a Dual Source scanner)
Period: Overall Study
Arm/Group | Myocardial Stress CT Perfusion Imaging
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Myocardial Stress CT Perfusion Imaging: Patients who will undergo myocardial stress CT perfusion imaging.
Arm/Group | Myocardial Stress CT Perfusion Imaging
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Per-Vessel Sensitivity of CTP in the Detection of Myocardial Perfusion Defects During Pharmacological Stress as Compared to Invasive Angiography.
Description: The gold standard for abnormality by CTP is defined as a focal stenosis of >50% at quantitative analysis of invasive coronary angiography images, when performed.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myocardial Stress CT Perfusion Imaging
Number analyzed (Participants) | 50
percentage of participants | 79 [63 to 90]

2. Secondary Outcome: Per-Patient Correlation Between CTP and SPECT at Stress.
Description: Pearson Correlation between research interpretation of CTP images and SPECT images, both performed during stress.
Time Frame: 18 months
Measure: Number; unit: correlation coefficient
Arm/Group | Myocardial Stress CT Perfusion Imaging
Number analyzed (Participants) | 50
correlation coefficient | 0.60
Statistical Analysis 1: Comparison: Myocardial Stress CT Perfusion Imaging; Test type: Superiority or Other; p < 0.0001, Pearson Correlation

3. Primary Outcome: Per-Vessel Specificity of CTP in the Detection of Myocardial Perfusion Defects During Pharmacological Stress as Compared to Invasive Angiography.
Description: The gold standard for abnormality by CTP is defined as stenosis of 50% or more at quantitative analysis of invasive coronary angiography images, when performed.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Myocardial Stress CT Perfusion Imaging
Number analyzed (Participants) | 50
percentage of participants | 80 [68 to 89]

4. Secondary Outcome: Per-Patient Correlation Between CTP and SPECT at Rest.
Description: Pearson Correlation performed on myocardial abnormalities on CTP and SPECT images, obtained at rest.
Time Frame: 18 months
Measure: Number; unit: correlation coefficient
Arm/Group | Myocardial Stress CT Perfusion Imaging
Number analyzed (Participants) | 50
correlation coefficient | 0.76
Statistical Analysis 1: Comparison: Myocardial Stress CT Perfusion Imaging; Pearson Correlation; Test type: Superiority or Other; p < 0.0001, Pearson Correlation

ADVERSE EVENTS:
Time Frame: 1 day
Description: To assure subject's safety, the study physician will monitor the safety of the subject. Heart rate and blood pressure will be measured immediately prior and 2 and 5 minutes after the administration of adenosine. ECG and heart rate will be continuously monitored during scanning. If adverse events occur the exam will immediately be stopped.
Arm/Group | Myocardial Stress CT Perfusion Imaging
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
Single-Center Study, Referral Population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less